CLINICAL TRIAL: NCT01792466
Title: A Randomized Controlled Trial of the Double Wire Technique With or Without Transpancreatic Sphincterotomy for Difficult Common Bile Duct Cannulation
Brief Title: RCT of the Double Wire Technique for Sphincterotomy
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Inadequate recruitment
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Douglas O. Faigel, Gastroenterologist, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 12-007021
Record Dates: First submitted 2013-02-11; First posted 2013-02-15 (Estimated); Last update posted 2017-07-21 (Actual); Status verified 2017-07

CONDITIONS: Cholangiopancreatography, Endoscopic Retrograde; Sphincterotomy, Endoscopic; VATER'S AMPULLA
Keywords: difficult biliary cannulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Transpacnreatic sphincterotomy (Experimental): In patients randomized to TPS, a transpancreatic sphincterotomy will be performed with the sphincterotome superficially in the pancreatic duct over a wire.
  Interventions: Procedure: Transpancreatic sphincterotomy
- Double wire without sphincterotomy (No Intervention): In patients randomized to the DWT group, the PD wire will be left in place, the catheter removed and then reinserted next to the PD wire with a second wire to attempt CBD cannluation

INTERVENTIONS:
Procedure: Transpancreatic sphincterotomy — A sphinctertome will be placed into the pancreatic duct over a guidewire and the sphincter will be cut in the direction of the bile duct
  Arms: Transpacnreatic sphincterotomy

SUMMARY:
Endoscopic cholangiography is a procedure which is performed to image the bile duct and perform therapy like removal of bile duct stones. It is currently standard of care to remove stones from the bile duct when found as they frequently cause complications like infections which can sometime be life threatening.

Therapy on the biliary tree, like for example stone removal, frequently requires inserting tools through the opening of the duct and cutting of the muscle which control the secretion of juices from the liver. Cutting the muscle helps with securing an easy access to the bile duct. It also helps facilitating dragging the stones out. On certain occasions placing a wire in the bile duct fails and instead the wire keeps entering the pancreatic duct whose opening is adjacent to the bile duct opening. There is evidence to suggest that keeping a wire in the pancreatic duct facilitates placing a second wire in the bile duct possibly because it straightens the duct. On certain occasions this also fails and we resort to cutting the muscle of the pancreas and the bile duct simultaneously to facilitate the access to the bile duct. The more attempt to enter the bile duct the higher the risk of inflammation in the pancreas known as pancreatitis. This makes decreasing the number of attempts at placing the wire in the duct desirable. One way to facilitate placement of the wire in the bile duct is to cut starting from the opening of the pancreas duct aiming toward the bile duct muscle. This often cuts the bile duct sphincter and exposes the bile duct opening. The study is trying to answer if cutting the bile duct sphincter muscle in the direction of the bile duct immediately after a wire has entered the pancreatic duct will make it easier to place the wire in the bile duct as compared to trying to place the wire in the bile duct without cutting the opening. While cutting the muscle canincrease the risk of pancreatitis, repeated attempts at accessing the bile duct can also increase the risk of pancreatitis. So if cutting the pancreatic muscle will facilitate entry to the bile duct and decrease the number of attempts at entering the bile duct then it might be a better way to approach the patient whom we had difficulty in entering the bile duct.

DETAILED DESCRIPTION:
This will be a prospective, non blinded randomized controlled trial. We will screen and offer enrollment to all patients presenting to Mayo Clinic Arizona for an ERCP who have a native papilla and an indication for cholangiography and sphincterotomy. Informed consent will be obtained in the preoperative area after obtaining consent for the ERCP. We will randomize all patients in whom we fail to deeply cannulate the CBD using a sphincterotome (Autotome, Boston Scientific) and 0.035" guidewire (0.035" Jagwire or Dreamwire, Boston Scientific) in over 5 minutes or with more than 5 attempts and in whom the wire can be passed in a stable configuration in the Pancreatic duct (PD). We will exclude patients who have any contraindication to undergoing an ERCP, contraindications to sphincterotomy (e,g,, abnormal anatomy, uncorrectable coagulopathy) and those who have pancreas divisum. Patients will be randomized 1:1 using opaque envelopes in blocks of 4 stratified for gender. (Gender stratification is necessary as the risks of ERCP vis pancreatitis are different for males and females). In those randomized to the DWT group, the PD wire will be left in place, the catheter removed and then reinserted next to the PD wire with a second wire to attempt CBD cannluation as previously described (1). In those randomized to TPS, a pancreatic sphincterotomy will be performed with the sphincterotome. The catheter will be removed with the PD wire left in place. The catheter and a second wire will be inserted and CBD cannluation attempted as for the DWT group. All patients will receive a 5Fr pancreatic stent and indomethacin 100 mg rectally to reduce the risk of pancreatitis as per our standard of care (patients with contraindications to NSAIDs (e.g., sensitivity to Indomethacin, aspirin or class, active peptic ulcer disease) will not receive Indomethacin. Patients who fail DWT (at least 10 minutes or 10 further attempts) may be crossed over to TPS at the endoscopist's discretion. Further care the patients receive will be standard of care. We will contact the patients around a months later by telephone to ask about any procedure related complications that were not reported to us.

outcome measures will be assessed on day 1 at the end of the procedure and on day 30.

ELIGIBILITY:
Inclusion criteria

1. All patients presenting to Mayo Clinic Arizona for an ERCP who have a native papilla
2. Failure to deeply cannulate the CBD in over 5 minutes and with more than 5 attempts
3. Stable wire placement into the Pancreatic duct (PD) exclusion criteria

1. Any contraindication to undergoing an ERCP. 2. Contraindications to sphincterotomy. 3. Pancreas divisum.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2013-02; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Number of attempts needed to achieve deep cannulation with a second wire. | Day one
  Number of attempts needed to achieve deep cannulation with a second wire.

SECONDARY OUTCOMES:
Time from randomization to deep cannulation. | day of the procedure
  Time from wire stable in the pancreatic duct until the second wire enters the bile duct

CONTACTS AND LOCATIONS:
Overall Officials: Douglas Faigel, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Arizona, Scottsdale, Arizona, United States